CLINICAL TRIAL: NCT02069158
Title: DOSE FINDING STUDY OF PF-05212384 WITH PACLITAXEL AND CARBOPLATIN IN PATIENTS WITH ADVANCED SOLID TUMOR
Acronym: IOSI-NDU-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cristiana Sessa (Other)
Responsible Party: Sponsor-Investigator, Cristiana Sessa, Prof., Oncology Institute of Southern Switzerland
Organization: Oncology Institute of Southern Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOSI-NDU-001
Record Dates: First submitted 2014-02-12; First posted 2014-02-24 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer; NSCLC; Ovary Cancer; Endometrial Cancer; Small Cell Lung Cancer (SCLC); Head and Neck (HNSCC)
Keywords: Advanced solid tumor
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Small Cell Lung Carcinoma; Squamous Cell Carcinoma of Head and Neck | interventions — gedatolisib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-05212384, Carboplatin, Paclitaxel (Experimental): starting dose of PF-05212384: 95 mg iv weekly Dose of Carboplatin: 5 AUC every 28 days Dose of Paclitaxel: 80 mg/m2 on days 1, 8 and 15
  Interventions: Drug: PF-05212384; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: PF-05212384 — iv administrartion
Drug: Paclitaxel — iv administration
  Other Names: Taxol
Drug: Carboplatin — iv administration
  Other Names: no applicable

SUMMARY:
This is a phase Ib single arm, open-label, multiple dose, dose escalating, safety, pharmacokinetic and pharmacodynamic study of the combination of PF-05212384 with paclitaxel and carboplatin. The study will be conducted in adult patients with advanced breast, NSCLC, ovarian or endometrial, small cell lung cancer (SCLC) and Head and Neck (HNSCC) cancer for whom there is an indication to the use of paclitaxel and carboplatin.

Successive cohorts of patients will receive escalating doses of PF-05212384 in combination with paclitaxel and carboplatin, starting at a dose level determined to be the 60% of single agent MTD.

The study will consist of two parts: the dose finding part (Part 1) and the expansion part (Part 2).

During Part 1 patients with breast, NSCLC, ovary and endometrial, small cell lung cancer (SCLC) and Head and Neck (HNSCC) cancer will be enrolled.

During Part 2, only patients with ovarian cancer will be enrolled. In Part 1, a 3+3 design is employed. Once the MTD of the combination is defined in Part 1, Part 2 is performed for a better definition of the safety profile, of the potential antitumor activity and of the pharmacodynamic effects of the combination; it will be conducted in at least 12 patients with ovarian cancer.

Approximately 40 patients are expected to be enrolled in the study overall.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Histological or cytological diagnosis of advanced/metastatic breast, NSCLC, ovarian and endometrial, small cell lung cancer (SCLC) and Head and Neck (HNSCC) cancer for which there is an indication to the use of paclitaxel and carboplatin.
* For patients enrolled to Part 1, lesions may be measurable or non measurable; for patients enrolled to Part 2, at least one measurable lesion is requested.
* All patients must provide an archived or fresh tumor sample; paired fresh tumor biopsies are mandatory for patients enrolled to Part 2 (at baseline and on Day 22 of Cycle 1).
* ECOG Performance Status must be 0 or 1.
* Adequate Bone Marrow Function, including:

  1. Absolute Neutrophil Count (ANC) ≥1,500/mm3 (or ≥1.5 x 109/L);
  2. Platelets ≥100,000/mm3 (or ≥100 x 109/L);
  3. Hemoglobin ≥9 g/dL.
* Adequate renal function, including: serum creatinine ≤1.5 x upper limit of normal (ULN) or estimated creatinine clearance ≥ 60 ml/min as calculated using the method standard for the institution.
* Adequate Liver Function, including:

  1. Total serum bilirubin ≤1.0 mg/dL Aspartate and Alanine Aminotransferase AST & ALT) ≤2.5 x ULN; ≤5.0 x ULN if there is liver involvement secondary to tumor.
  2. Alkaline phosphatase ≤2.5 x ULN; (≤5 x ULN in case of bone metastasis).
* Adequate glucose control, including no previous diagnosis of diabetes mellitus and HbA1c <7%.
* Adequate cardiac function, including: 12 Lead ECG with normal tracing or non clinically significant changes that do not require medical intervention.
* Resolved acute effects of any prior therapy to baseline severity or Grade

  * 1 CTCAE except for AEs not constituting a safety risk by Investigator judgment.
* Serum/urine pregnancy test (for females of childbearing potential) negative at screening and at baseline.
* Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. Male patients must be surgically sterile or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. The decision of effective contraception will be based on the judgment of the principal Investigator or a designated associate.
* Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.
* Written informed consent.

Exclusion Criteria:

* More than 2 prior lines of chemotherapy for advanced disease for Part 1, more than 1 prior line of chemotherapy for advanced disease for Part 2.
* Resistance to platinum agents (progression during the treatment or within 3 month from the stop of the treatment).
* Prior treatment with weekly paclitaxel with tumor progression.
* Pre-existing neuropathy ≥ G2.
* Patients with known active brain metastases. Patients with previously diagnosed brain metastases are eligible if they have completed their CNS treatment and have recovered from the acute effects of radiation therapy or surgery prior to the start of study medication, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable.
* Chemotherapy, radiotherapy (other than palliative radiotherapy to lesions that will not be followed for tumor assessment on this study, ie, non target lesions), biological or investigational agents within 4 weeks of the start of the study treatment (6 weeks for mitomycin C or nitrosoureas).
* Any surgery (not including minor procedures such as lymph node biopsy, needle biopsy, and/or placement of port-a-cath) within 4 weeks of the start of the study treatment or not fully recovered from any side effects of previous procedures.
* For patients enrolling to Part 2, prior therapy with an agent that is known or proposed to be active by action on PI3K and/or mTOR completed within the last 6 months.
* Uncontrolled or significant cardiovascular disease:
* A myocardial infarction within 12 months.
* Uncontrolled angina within 6 months.
* Congestive heart failure within 6 months.
* Diagnosed or suspected congenital long QT syndrome.
* Any history of ventricular arrhythmias (such as ventricular tachycardia, ventricular Fibrillation, or Torsades de pointes).
* Any history of second or third degree heart block (may be eligible if currently have a pacemaker).
* Heart rate <50/minute on pre entry electrocardiogram.
* Uncontrolled hypertension.
* Current use or anticipated need for food or drugs that are known potent CYP3A4 inhibitors. Because inhibition of CYP3A4 isoenzymes may increase PF- 05212384 exposure leading to a potential increases in toxicities, the use of known strong inhibitors (strong CYP3A4 Inhibitors: grapefruit juice or grapefruit/grapefruit related citrus fruits (eg, Seville oranges, pomelos), ketoconazole, miconazole, itraconazole, voriconazole, posaconazole, erythromycin, clarithromycin, telithromycin, verapamil, indinavir, saquinavir, ritonavir, nelfinavir, nefazodone, lopinavir, atazanavir, amprenavir, fosamprenavir and delavirdine, troleandomycin, mibefradil, conivaptan) are not permitted from 10 days prior to the first dose of study drug until discontinuation. Concurrent administration of herbal preparations and current or anticipated need for food or drugs that are known substrates of UGT1A9 (eg, propofol, acetaminophen, and propranolol), of which PF-05212384 is a strong inhibitor, is not permitted from 10 days prior to the first dose of study drug until discontinuation.
* Current or anticipated need for food or drugs that are known potent CYP3A4 inducers. PF-05212384 metabolism may be induced when taking strong CYP3A4 inducers (eg, phenobarbital, rifampin, phenytoin, carbamazepine, rifabutin, rifapentin, clevidipine, St. John's Wort) resulting in reduced plasma concentrations. Therefore co administration of study drug in combination with these and other strong CYP3A4 inducers is not permitted from 10 days prior to the first dose of study drug until study treatment discontinuation.
* Breast feeding or intercurrent pregnancy; no use of highly effective contraception or not agreeing to continue highly effective contraception for 90 days after last dose of investigational product.
* Any mental disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
dose limiting toxicity (DLT) | 28 days after the first administration
  Assessment of the dose limiting toxicities (DLT) during first cycle
Adverse Events | minimum 8 weeks
  Adverse Event characterized by type, frequency and severity (as graded by NCICTCAE v. 4.03) during the treatment until progessive disease
laboratory Adverse Events | minimum 8 weeks
  Laboratory abnormalities characterized by type, frequency and severity (as graded by NCICTCAE v. 4.03) during all treatment until progressive disease

SECONDARY OUTCOMES:
Pharmacokintecs of PF-05212384 | Cycle 1 day 1 and Cycle 2 day 1
  Evaluation of the pharmacokinetic of PF-05212384 single agent or in combination with paclitaxel and carboplatin
Tumor response | every 8 weeks
  Objective tumor response assessed by Response Evaluation Criteria in Solid Tumors (RECIST), RR, TTP
biomarkers of pathway inhibition | Day 1 of each cycle
  Serum glucose, and other circulating biomarkers of pathway inhibition (pS6K1)
Pharmacodynamic | Just before the treatment starts and cycle 1 day 22
  Evaluation of the pharmacodynamic of biomarkers in tumor tissues (archived and fresh tumor biopsy)
Gene expression | Just before the treatment starts
  Gene expression in biopsied tumor tissues (fresh or archived) relating to PI3K and MAPK signaling

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios Stathis, Prof., Principal Investigator — IOSI Sponsor Unit
Locations (1):
- Oncology Institute of Southern Switzerland (IOSI), Bellinzona, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No